CLINICAL TRIAL: NCT00553475
Title: Randomized, Double-Blind, Multicenter, Placebo-Controlled Study To Evaluate Efficacy And Safety Of Pregabalin (CI-1008) In The Treatment For Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Randomized, Double-Blind, Multicenter, Placebo-Controlled Study Of Pregabalin For Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081163
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2010-07

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Pregabalin 300 mg/day (Experimental)
  Interventions: Drug: pregabalin
- Pregabalin 600 mg/day (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: placebo — Dosage: placebo, oral administration, Treatment duration: 13 weeks (1-week titration and 12-week fixed dose)
  Arms: Placebo
Drug: pregabalin — Dosage: 300 mg/day (150 mg bid), oral administration, Treatment duration: 13 weeks (1-week titration and 12-week fixed dose)
  Arms: Pregabalin 300 mg/day
Drug: pregabalin — Dosage: 600 mg/day (300 mg bid), oral administration, Treatment duration: 13 weeks (1-week titration and 12-week fixed dose)
  Arms: Pregabalin 600 mg/day

SUMMARY:
To evaluate the efficacy and safety of pregabalin at 300 mg/day and 600 mg/day (BID) in patients with painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Visual Analogue Scale (VAS) of pain is higher than 40 mm.
* Diagnosis of type 1 or 2 diabetes mellitus for at least 1 year

Exclusion Criteria:

* Malignancy within the past 2 years.
* Neurologic disorders unrelated to diabetic neuropathy that may confuse the assessment of neuropathy pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- Japan (49):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chikushino-shi, Fukuoka
  - Pfizer Investigational Site, Kasuga, Fukuoka
  - Pfizer Investigational Site, Date-shi, Fukushima
  - Pfizer Investigational Site, Nihommatsu, Fukushima
  - Pfizer Investigational Site, Shirakawa-shi, Fukushima
  - Pfizer Investigational Site, Sukagawa, Fukushima
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Chitose, Hokkaido
  - Pfizer Investigational Site, Ebetu, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaiido
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Inashiki, Ibaraki
  - Pfizer Investigational Site, Kamakura, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Yatsushiro, Kumamoto
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Matsumoto, Nagano
  - Pfizer Investigational Site, Ueda, Nagano
  - Pfizer Investigational Site, Beppu, Oita Prefecture
  - Pfizer Investigational Site, Yamada, Okayama-ken
  - Pfizer Investigational Site, Naha, Okinawa
  - Pfizer Investigational Site, Tomishiro, Okinawa
  - Pfizer Investigational Site, Urazoe, Okinawa
  - Pfizer Investigational Site, Higashiosaka, Osaka
  - Pfizer Investigational Site, Hirano-ku, Osaka
  - Pfizer Investigational Site, Kishiwada, Osaka
  - Pfizer Investigational Site, Suminoe-ku, Osaka
  - Pfizer Investigational Site, Sunto-gun, Shizuoka
  - Pfizer Investigational Site, Oyama-shi, Tochigi
  - Pfizer Investigational Site, Utsunomiya, Tochigi
  - Pfizer Investigational Site, Arakawa City, Tokyo
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Chuo-ku, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Nishitōkyō, Tokyo
  - Pfizer Investigational Site, Ohta-ku, Tokyo
  - Pfizer Investigational Site, Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Kumamoto
  - Pfizer Investigational Site, Nagasaki
  - Pfizer Investigational Site, Niigata
  - Pfizer Investigational Site, Okayama
  - Pfizer Investigational Site, Ōita
  - Pfizer Investigational Site, Saga
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Tokushima

REFERENCES:
- [Derived] Alexander J Jr, Edwards RA, Manca L, Grugni R, Bonfanti G, Emir B, Whalen E, Watt S, Brodsky M, Parsons B. Integrating Machine Learning With Microsimulation to Classify Hypothetical, Novel Patients for Predicting Pregabalin Treatment Response Based on Observational and Randomized Data in Patients With Painful Diabetic Peripheral Neuropathy. Pragmat Obs Res. 2019 Oct 31;10:67-76. doi: 10.2147/POR.S214412. eCollection 2019. PMID 31802967
- [Derived] Alexander J Jr, Edwards RA, Brodsky M, Manca L, Grugni R, Savoldelli A, Bonfanti G, Emir B, Whalen E, Watt S, Parsons B. Using time series analysis approaches for improved prediction of pain outcomes in subgroups of patients with painful diabetic peripheral neuropathy. PLoS One. 2018 Dec 6;13(12):e0207120. doi: 10.1371/journal.pone.0207120. eCollection 2018. PMID 30521533
- [Derived] Edwards RA, Bonfanti G, Grugni R, Manca L, Parsons B, Alexander J. Predicting Responses to Pregabalin for Painful Diabetic Peripheral Neuropathy Based on Trajectory-Focused Patient Profiles Derived from the First 4 Weeks of Treatment. Adv Ther. 2018 Oct;35(10):1585-1597. doi: 10.1007/s12325-018-0780-3. Epub 2018 Sep 11. PMID 30206821
- [Derived] Parsons B, Li C, Emir B, Vinik AI. The efficacy of pregabalin for treating pain associated with diabetic peripheral neuropathy in subjects with type 1 or type 2 diabetes mellitus. Curr Med Res Opin. 2018 Nov;34(11):2015-2022. doi: 10.1080/03007995.2018.1509304. Epub 2018 Sep 20. PMID 30084288
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081163&StudyName=Randomized%2C%20Double-Blind%2C%20Multicenter%2C%20Placebo-Controlled%20Study%20Of%20Pregabalin%20For%20Pain%20Associated%20With%20Diabetic%20Peripheral%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 1-week baseline phase, subjects were classified into 2 strata based on creatinine clearance (CLcr) values (Low: 30 <CLcr <=60 mL/minute; Normal: CLcr > 60 mL/minute) and were each randomly assigned to 1 of 3 treatment groups.
Groups:
- Placebo: During a 13-week double-blind phase, subjects received matching placebo.
- Pregabalin 300 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects received pregabalin 300 mg/day for 12 weeks.
- Pregabalin 600 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects with low CLcr received pregabalin 300 mg/day and subjects with normal CLcr received pregabalin 600 mg/day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Started | 135 | 134 | 45
Completed | 119 | 114 | 32
Not Completed | 16 | 20 | 13
Not completed — Adverse Event | 7 | 17 | 13
Not completed — Lack of Efficacy | 7 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Due to moving | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day | Total
Number analyzed (Participants) | 135 | 134 | 45 | 314
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0 | 0
  18 - 44 years | 7 | 8 | 1 | 16
  45 - 64 years | 76 | 78 | 25 | 179
  >= 65 years | 52 | 48 | 19 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.6) | 61.3 (10.3) | 62.2 (10.3) | 61.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 13 | 77
  Male | 103 | 102 | 32 | 237
Region of Enrollment [Number; unit: participants]
  Japan | 135 | 134 | 45 | 314

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Study Endpoint in Mean Weekly Pain Scores
Description: Change from baseline: Score at study endpoint minus score at baseline. Study endpoint is defined as the mean of the last seven entries of the daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) while on study medication up to and including day after last dose.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -1.20 (0.21) | -1.82 (0.22) | -1.94 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0075, ANCOVA; Treatment groups and the CLcr strata as factors and baseline values as covariates; Mean Difference (Final Values) = -0.63, 95% CI [-1.09 to -0.17]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0254, ANCOVA; Treatment groups and the CLcr strata as factors and baseline values as covariates; Mean Difference (Final Values) = -0.74, 95% CI [-1.39 to -0.09]

2. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Physical Functioning
Description: The mean change from baseline in Short-Form 36-Item Health Survey Scores at study endpoint. Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 2.70 (1.58) | 2.43 (1.59) | 3.86 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.8731, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.28, 95% CI [-3.67 to 3.12]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.6337, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.16, 95% CI [-3.62 to 5.94]

3. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Role Limitations-Physical
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 4.38 (2.47) | 2.28 (2.50) | 3.97 (3.70)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4398, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.10, 95% CI [-7.44 to 3.24]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.9153, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.41, 95% CI [-7.96 to 7.14]

4. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Bodily Pain
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 10.34 (1.97) | 11.84 (1.99) | 12.89 (2.91)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4873, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.50, 95% CI [-2.75 to 5.76]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4008, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 2.56, 95% CI [-3.42 to 8.53]

5. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: General Health Perception
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 2.31 (1.44) | 3.29 (1.45) | 4.40 (2.14)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.5372, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.98, 95% CI [-2.13 to 4.09]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.3480, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 2.09, 95% CI [-2.29 to 6.47]

6. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Social Functioning
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 3.00 (2.39) | 8.06 (2.41) | 11.16 (3.54)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0544, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.06, 95% CI [-0.10 to 10.21]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0278, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 8.15, 95% CI [0.89 to 15.42]

7. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Role Limitations-Emotional
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 4.13 (2.52) | 5.05 (2.55) | 6.35 (3.77)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.7394, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.92, 95% CI [-4.52 to 6.37]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.5712, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 2.22, 95% CI [-5.49 to 9.93]

8. Primary Outcome: Change From Baseline to Study Endpoint in Mean Weekly Pain Scores by Groups of Subjects With Expected Similar Plasma Concentrations
Description: Change from baseline: Score at study endpoint minus score at baseline. Study endpoint is defined as the mean of the last seven entries of the daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) while on study medication up to and including day after last dose. Subjects are classified by exposure to pregabalin, which is estimated by creatinine clearance (CLcr).
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Groups:
- Expected Exposure Pregabalin 300 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects with normal CLcr in the pregabalin 300 mg/day group received pregabalin 300 mg/day for 12 weeks.
- Expected Exposure Pregabalin 600 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects with low CLcr in the pregabalin 300 and 600 mg/day groups received pregabalin 300 mg/day and subjects with normal CLcr in the pregabalin 600 mg/day group received pregabalin 600 mg/day for 12 weeks.
Arm/Group | Placebo | Expected Exposure Pregabalin 300 mg/Day | Expected Exposure Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 120 | 59
score on scale | -1.27 (0.16) | -1.93 (0.17) | -1.90 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Expected Exposure Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0058, ANCOVA; Treatment groups as factors and baseline values as covariates; Mean Difference (Final Values) = -0.67, 95% CI [-1.14 to -0.19]
Statistical Analysis 2: Comparison: Placebo vs Expected Exposure Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0333, ANCOVA; Treatment groups as factors and baseline values as covariates; Mean Difference (Final Values) = -0.64, 95% CI [-1.23 to -0.05]

9. Primary Outcome: Number of Responders
Description: A responder is defined as a subject with a 50% reduction in weekly mean pain score from baseline to study endpoint.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
participants | 29 | 39 | 16
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Significance level of 0.05 was used; Test type: Superiority or Other; p = 0.153, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Significance level of 0.05 was used; Test type: Superiority or Other; p = 0.059, Cochran-Mantel-Haenszel; stratified by CLcr stratum

10. Primary Outcome: Change From Baseline at Week 1 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 1.
  Change from baseline: Score at Week 1 minus score at baseline
Time Frame: From baseline to Week 1
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -0.39 (0.17) | -0.82 (0.17) | -1.14 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0287, Mixed Model Repeated Measures Analysis; Model included treatment, CLcr stratum, week and treatment-by-week interaction, and baseline scores as fixed effects, and subject as a random effect; Mean Difference (Final Values) = -0.43, 95% CI [-0.82 to -0.05]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0073, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Median Difference (Final Values) = -0.75, 95% CI [-1.29 to -0.20]

11. Primary Outcome: Change From Baseline at Week 2 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 2.
  Change from baseline: Score at Week 2 minus score at baseline
Time Frame: From baseline to Week 2
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 133 | 132 | 41
score on scale | -0.57 (0.17) | -1.17 (0.17) | -1.80 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0021, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI [-1.00 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.23, 95% CI [-1.78 to -0.69]

12. Primary Outcome: Change From Baseline at Week 3 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 3.
  Change from baseline: Score at Week 3 minus score at baseline
Time Frame: From baseline to Week 3
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 131 | 129 | 41
score on scale | -0.80 (0.17) | -1.40 (0.17) | -1.93 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0026, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.60, 95% CI [-0.99 to -0.21]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.13, 95% CI [-1.69 to -0.58]

13. Primary Outcome: Change From Baseline at Week 4 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 4.
  Change from baseline: Score at Week 4 minus score at baseline
Time Frame: From baseline to Week 4
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 130 | 128 | 41
score on scale | -0.89 (0.17) | -1.53 (0.17) | -2.00 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0012, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI [-1.03 to -0.25]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.11, 95% CI [-1.67 to -0.56]

14. Primary Outcome: Change From Baseline at Week 5 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 5.
  Change from baseline: Score at Week 5 minus score at baseline
Time Frame: From baseline to Week 5
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 130 | 125 | 38
score on scale | -0.91 (0.17) | -1.57 (0.17) | -2.07 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0011, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI [-1.04 to -0.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.16, 95% CI [-1.72 to -0.60]

15. Primary Outcome: Change From Baseline at Week 6 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 6.
  Change from baseline: Score at Week 6 minus score at baseline
Time Frame: From baseline to Week 6
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 128 | 125 | 37
score on scale | -0.94 (0.17) | -1.72 (0.17) | -2.06 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.79, 95% CI [-1.18 to -0.40]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.12, 95% CI [-1.68 to -0.56]

16. Primary Outcome: Change From Baseline at Week 7 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 7.
  Change from baseline: Score at Week 7 minus score at baseline
Time Frame: From baseline to Week 7
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 125 | 124 | 36
score on scale | -1.04 (0.17) | -1.76 (0.17) | -2.13 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0003, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.72, 95% CI [-1.12 to -0.33]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0002, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -1.09, 95% CI [-1.66 to -0.52]

17. Primary Outcome: Change From Baseline at Week 8 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 8.
  Change from baseline: Score at Week 8 minus score at baseline
Time Frame: From baseline to Week 8
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 125 | 123 | 36
score on scale | -1.18 (0.17) | -1.85 (0.17) | -2.12 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0008, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.67, 95% CI [-1.07 to -0.28]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0014, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.94, 95% CI [-1.51 to -0.36]

18. Primary Outcome: Change From Baseline at Week 9 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 9.
  Change from baseline: Score at Week 9 minus score at baseline
Time Frame: From baseline to Week 9
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 123 | 121 | 35
score on scale | -1.20 (0.17) | -1.93 (0.17) | -2.06 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0003, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.73, 95% CI [-1.12 to -0.33]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0036, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI [-1.44 to -0.28]

19. Primary Outcome: Change From Baseline at Week 10 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 10.
  Change from baseline: Score at Week 10 minus score at baseline
Time Frame: From baseline to Week 10
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 122 | 118 | 33
score on scale | -1.23 (0.17) | -1.93 (0.18) | -2.10 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0005, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI [-1.10 to -0.31]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0034, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI [-1.46 to -0.29]

20. Primary Outcome: Change From Baseline at Week 11 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 11.
  Change from baseline: Score at Week 11 minus score at baseline
Time Frame: From baseline to Week 11
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 121 | 116 | 33
score on scale | -1.32 (0.17) | -1.95 (0.18) | -2.09 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0023, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI [-1.02 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0105, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI [-1.36 to -0.18]

21. Primary Outcome: Change From Baseline at Week 12 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 12.
  Change from baseline: Score at Week 12 minus score at baseline
Time Frame: From baseline to Week 12
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 120 | 116 | 33
score on scale | -1.36 (0.17) | -2.01 (0.18) | -2.13 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0016, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI [-1.05 to -0.25]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0111, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI [-1.37 to -0.18]

22. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Vitality
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 5.28 (1.92) | 4.20 (1.94) | 12.87 (2.84)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.6118, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.07, 95% CI [-5.23 to 3.08]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0109, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 7.59, 95% CI [1.76 to 13.42]

23. Secondary Outcome: Change From Baseline in Short Form 36-Item (SF-36) Health Survey: Mental Health
Description: as for outcome 2
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 3.84 (1.83) | 5.33 (1.85) | 7.81 (2.72)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4602, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.49, 95% CI [-2.47 to 5.45]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1625, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.97, 95% CI [-1.61 to 9.54]

24. Secondary Outcome: Change From Baseline in Mean Sleep Interference Scores
Description: The mean change from baseline in the weekly mean sleep interference score at study endpoint. Score range is from 0-10. Higher scores indicate more severe interference with sleep.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -0.74 (0.18) | -1.59 (0.18) | -1.36 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.85, 95% CI [-1.25 to -0.46]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0273, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.63, 95% CI [-1.19 to -0.07]

25. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Sensory Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Sensory score ranges from 0-33. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -2.82 (0.50) | -4.60 (0.50) | -4.95 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0013, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.79, 95% CI [-2.87 to -0.71]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0062, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.13, 95% CI [-3.65 to -0.61]

26. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Affective Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Affective score ranges from 0-12. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -0.83 (0.20) | -1.43 (0.20) | -1.39 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0068, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.60, 95% CI [-1.03 to -0.17]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0707, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.56, 95% CI [-1.17 to 0.05]

27. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Total Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Total score ranges from 0-45. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -3.68 (0.66) | -6.03 (0.66) | -6.36 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0013, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.35, 95% CI [-3.76 to -0.93]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0087, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.67, 95% CI [-4.67 to -0.68]

28. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Visual Analogue Scale Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Visual Analogue Scale Score ranges from 0-100 mm. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
mm | -16.92 (2.38) | -24.19 (2.40) | -24.41 (3.53)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0056, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -7.27, 95% CI [-12.40 to -2.14]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0427, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -7.49, 95% CI [-14.74 to -0.25]

29. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Present Pain Intensity Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Present pain intensity score ranges from 0-5. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 134 | 45
score on scale | -0.59 (0.09) | -0.80 (0.09) | -0.96 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0365, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.21, 95% CI [-0.40 to -0.01]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0073, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.37, 95% CI [-0.65 to -0.10]

30. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Sleep Disturbance
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for sleep disturbance ranges from 0-100. Higher scores indicate more severe pain.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | -9.03 (1.86) | -15.40 (1.88) | -12.81 (2.77)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0019, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -6.37, 95% CI [-10.38 to -2.36]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1907, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -3.78, 95% CI [-9.45 to 1.89]

31. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Snoring
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for snoring ranges from 0-100. Higher scores indicate more of the attribute.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | -6.00 (2.51) | -5.96 (2.53) | -1.56 (3.71)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.9905, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.03, 95% CI [-5.37 to 5.43]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.2532, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 4.44, 95% CI [-3.19 to 12.08]

32. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Sleep Shortness of Breath or Headache
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for sleep shortness of breath or headache ranges from 0-100. Higher scores indicate more of the attribute.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | -1.63 (1.69) | -3.02 (1.71) | -4.47 (2.51)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4538, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.39, 95% CI [-5.05 to 2.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.2782, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.84, 95% CI [-7.97 to 2.30]

33. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Quantity of Sleep
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for quantity of sleep ranges from 0-24. Higher scores indicate more of the attribute named in the subscale.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 0.37 (0.12) | 0.69 (0.12) | 0.54 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0177, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.32, 95% CI [0.06 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.3661, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.17, 95% CI [-0.20 to 0.55]

34. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Sleep Adequacy
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for sleep adequacy ranges from 0-100. Higher scores indicate more of the attribute.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 12.08 (2.61) | 17.69 (2.64) | 21.73 (3.87)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0511, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.62, 95% CI [-0.03 to 11.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0173, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 9.65, 95% CI [1.72 to 17.59]

35. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Somnolence
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for somnolence ranges from 0-100. Higher scores indicate more of the attribute.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 134 | 133 | 45
score on scale | -2.96 (2.17) | 0.83 (2.19) | 4.83 (3.20)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1123, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.79, 95% CI [-0.89 to 8.47]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0206, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 7.79, 95% CI [1.20 to 14.38]

36. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) - Sleep Scale: Overall Sleep Problems Index
Description: The mean change from baseline in Medical Outcomes Study - Sleep Scale Scores at study endpoint. Score for overall sleep problems index ranges from 0-100. Higher scores indicate more of the attribute.
Time Frame: From baseline to Week 13 or up to study discontinuation (Study Endpoint)
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | -7.91 (1.45) | -11.45 (1.46) | -9.73 (2.16)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0269, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -3.54, 95% CI [-6.67 to -0.41]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.4183, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.82, 95% CI [-6.24 to 2.60]

37. Secondary Outcome: Clinical Global Impression of Change
Description: Clinical Global Impression of Change is a clinician-rated instrument that measures change in patient's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 13 or up to discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 3.3 (1.2) | 2.9 (1.1) | 2.7 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0148, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi-squared with a modified ridit transformation, stratified by stratum based on the CLcr
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi-squared with a modified ridit transformation, stratified by stratum based on the CLcr

38. Secondary Outcome: Patient Global Impression of Change
Description: The Patient Global Impression of Change is a patient-rated instrument that measures change in patient's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 13 or up to discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 135 | 133 | 45
score on scale | 3.4 (1.3) | 3.2 (1.0) | 2.8 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0818, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi-squared with a modified ridit transformation, stratified by stratum based on the CLcr
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0075, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi-squared with a modified ridit transformation, stratified by stratum based on the CLcr

39. Primary Outcome: Change From Baseline at Week 13 in Mean Weekly Pain Scores
Description: The mean change from baseline in mean weekly pain score from daily pain diary using the 11-point numerical rating scale 0(no pain) to 10(worst possible pain) at Week 13.
  Change from baseline: Score at Week 13 minus score at baseline
Time Frame: From baseline to Week 13
Population: Full analysis set. Observed case (No imputation).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 119 | 115 | 33
score on scale | -1.38 (0.17) | -2.04 (0.18) | -2.12 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0013, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.66, 95% CI [-1.07 to -0.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0152, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.74, 95% CI [-1.34 to -0.14]

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Serious Adverse Events (participants affected / at risk) | 3/135 | 2/134 | 1/45
Other Adverse Events (participants affected / at risk) | 50/135 | 71/134 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=135) | Pregabalin 300 mg/Day (N=134) | Pregabalin 600 mg/Day (N=45)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Peripheral coldness (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=135) | Pregabalin 300 mg/Day (N=134) | Pregabalin 600 mg/Day (N=45)
Constipation (Gastrointestinal disorders) | 1 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 3
Oedema (General disorders) | 1 | 4 | 3
Oedema peripheral (General disorders) | 8 | 19 | 8
Nasopharyngitis (Infections and infestations) | 20 | 16 | 4
Weight increased (Investigations) | 5 | 17 | 7
Dizziness (Nervous system disorders) | 9 | 26 | 18
Somnolence (Nervous system disorders) | 12 | 28 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.